CLINICAL TRIAL: NCT04065451
Title: Effect of Epinephrine on Immediate Post-polypectomy Pain in Colorectal Lesions Larger Than 20 mm
Brief Title: Effect of Epinephrine on Post-polypectomy Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Douglas K. Rex, Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1908473351
Record Dates: First submitted 2019-08-15; First posted 2019-08-22 (Actual); Results first posted 2022-09-30 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Colonic Polyp
MeSH Terms: conditions — Colonic Polyps | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Epinephrine (Experimental): Epinephrine in the submucosal injection fluid (1:200,000)
  Interventions: Drug: Epinephrine
- No epinephrine (No Intervention): Submucosal injection fluid without epinephrine

INTERVENTIONS:
Drug: Epinephrine — Epinephrine in the submucosal injection fluid
  Arms: Epinephrine

SUMMARY:
Epinephrine is widely used in endoscopic mucosal resection of large polyps to prevent post-polypectomy bleeding. No previous studies looked at increase in immediate post-polypectomy pain with the use of epinephrine.

ELIGIBILITY:
Inclusion Criteria

1. Patients aged 18 years and over
2. Patients scheduled for treatment of large (≥ 20 mm) colorectal polyps
3. Able to sign informed consent

Exclusion Criteria

1. Patients previously enrolled in the study
2. Pedunculated polyps
3. Polyps not amenable to endoscopic resection
4. Patients allergic or sensitive to epinephrine
5. Patients with coronary artery disease who have had a myocardial infarction in the past year, or had coronary stenting in the past year, or had angina in the past year.
6. Patients electing anesthesia other than monitored anesthesia care with propofol (MAC) for colonoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas K Rex, MD, Principal Investigator — IU
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pohl H, Srivastava A, Bensen SP, Anderson P, Rothstein RI, Gordon SR, Levy LC, Toor A, Mackenzie TA, Rosch T, Robertson DJ. Incomplete polyp resection during colonoscopy-results of the complete adenoma resection (CARE) study. Gastroenterology. 2013 Jan;144(1):74-80.e1. doi: 10.1053/j.gastro.2012.09.043. Epub 2012 Sep 25. PMID 23022496
- [Background] ASGE Technology Committee; Hwang JH, Konda V, Abu Dayyeh BK, Chauhan SS, Enestvedt BK, Fujii-Lau LL, Komanduri S, Maple JT, Murad FM, Pannala R, Thosani NC, Banerjee S. Endoscopic mucosal resection. Gastrointest Endosc. 2015 Aug;82(2):215-26. doi: 10.1016/j.gie.2015.05.001. Epub 2015 Jun 12. PMID 26077453
- [Background] Klein A, Bourke MJ. How to Perform High-Quality Endoscopic Mucosal Resection During Colonoscopy. Gastroenterology. 2017 Feb;152(3):466-471. doi: 10.1053/j.gastro.2016.12.029. Epub 2017 Jan 3. No abstract available. PMID 28061339
- [Background] World Health Organization. Epinephrine (for use with local anaesthetics). Model Prescribing Information: Drugs Used in Anaesthesis, Geneva, 1989:33
- [Derived] Rex DK, Lahr RE, Peterson MM, Vemulapalli KC. Impact of including epinephrine in the submucosal injectate for colorectal EMR on postprocedural pain: a randomized controlled trial. Gastrointest Endosc. 2022 Mar;95(3):535-539.e1. doi: 10.1016/j.gie.2021.11.043. Epub 2021 Dec 9. PMID 34896443

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty-two patients consented to participate in the trial, but two patients were not randomized to either of the study arms. One patient did not have a polyp to remove (referred polyp was a lipoma). The other patient had poor bowel preparation, and the procedure was aborted.
Period: Overall Study
Arm/Group | Epinephrine | No Epinephrine
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: Other Units (Polyps)
Groups:
- Total: Total of all reporting groups
Arm/Group | Epinephrine | No Epinephrine | Total
Number analyzed (Participants) | 10 | 10 | 20
Number analyzed (Other Units (Polyps)) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (9.1) | 60.5 (9.1) | 61.4 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 4 | 3 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8 | 6 | 14
  Unknown/Not Reported | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
Polyp Size [Mean (Standard Deviation); unit: millimeters] | 46.7 (28.3) | 40.4 (16.1) | 43.7 (23.0)

OUTCOME MEASURES:

1. Primary Outcome: Immediate Post-polypectomy Pain
Description: Pain related by the participant on a 0-100 visual analog scale; patients will be asked to mark their pain level on a straight vertical line 100 mm long and this point will be measured with a ruler for pain score. Possible values are zero- indicating no pain at all to 100-indicating worst imaginable pain
Time Frame: 30 minutes after the procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epinephrine | No Epinephrine
Number analyzed (Participants) | 10 | 10
units on a scale | 46.5 (32.4) | 13.6 (25.9)

2. Primary Outcome: Immediate Post Polypectomy Pain (1hour)
Description: as for outcome 1
Time Frame: 1 hour after procedure
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Epinephrine | No Epinephrine
Number analyzed (Participants) | 10 | 10
Units on a Scale | 44 (27.7) | 12.9 (27.8)

3. Secondary Outcome: en Bloc Resection
Description: Number of polyps removed en bloc (in 1 piece) vs number of polyps removed piecemeal (in more than 1 piece)
Time Frame: During the colonoscopy procedure, an average of 47.3 minutes
Population: One patient in the epinephrine group had two eligible polyps for the study so there ended up being 11 polyps in the epinephrine arm.
Measure: Number; unit: Polyps
Units Other Than Participants: Polyps
Arm/Group | Epinephrine | No Epinephrine
Number analyzed (Participants) | 10 | 10
Number analyzed (Polyps) | 11 | 10
Polyps
  En bloc removal | 0 | 0
  Piecemeal removal | 11 | 10

4. Secondary Outcome: Sydney Resection Quotient
Description: size of the polyp in mm divided by the number of pieces the polyps is removed in
Time Frame: During the colonoscopy procedure, an average of 47.3 minutes
Population: Only lesions removed by EMR with electrocautery (heat) are included.
Measure: Median (Inter-Quartile Range); unit: Ratio
Units Other Than Participants: Polyps
Arm/Group | Epinephrine | No Epinephrine
Number analyzed (Participants) | 7 | 9
Number analyzed (Polyps) | 7 | 9
Ratio | 5 [4.1 to 6.3] | 4.2 [3.1 to 5.6]

5. Secondary Outcome: Quality of the Mound
Description: Endoscopist impression of lift provided by the submucosal injection: excellent/adequate or insufficient. Excellent is the best rating and insufficient is the worst rating on this scale.
Time Frame: During the colonoscopy procedure, an average of 47.3 minutes
Population: as for outcome 3
Measure: Count of Units; unit: Polyps
Units Other Than Participants: Polyps
Arm/Group | Epinephrine | No Epinephrine
Number analyzed (Participants) | 10 | 10
Number analyzed (Polyps) | 11 | 10
Polyps
  Excellent/adequate | 9 | 8
  insufficient | 0 | 2
  Unknown | 2 | 0

6. Secondary Outcome: Frequency of Immediate Bleeding
Description: Number of polyps with intraprocedural bleeding during removal
Time Frame: During the colonoscopy procedure, an average of 47.3 minutes
Population: as for outcome 3
Measure: Count of Units; unit: Polyps
Units Other Than Participants: Polyps
Arm/Group | Epinephrine | No Epinephrine
Number analyzed (Participants) | 10 | 10
Number analyzed (Polyps) | 11 | 10
Polyps
  Bleeding | 2 | 4
  No bleeding | 9 | 6

ADVERSE EVENTS:
Time Frame: 30 days
Description: Patients were assessed for adverse events that occurred within 30 days after the procedure
Arm/Group | Epinephrine | No Epinephrine
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epinephrine (N=10) | No Epinephrine (N=10)
delayed bleeding (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
abdominal pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
* Number of patients in study was small but sample size calculation was performed prior to initiating the study.
* Study conducted by single experienced endoscopist which might limit generalizability.
* Blinding to the use of epinephrine proved to not be possible due to the blanching effect of epinephrine.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/51/NCT04065451/Prot_SAP_000.pdf